CLINICAL TRIAL: NCT05169879
Title: Influence of Early Coronal Flaring Upon Postoperative Pain Following Root Canal Treatment. A Randomized Clinical Trial
Brief Title: Influence of Early Coronal Flaring Upon Postoperative Pain After Root Canal Treatment
Acronym: flaring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba Elasfouri, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Endo 28-11-2021
Record Dates: First submitted 2021-11-28; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early acoronal flaring (Experimental): In group A, ProGlider PG (size 16, .02 taper) instrument with a length of 25 mm will be used to the working length, then early coronal flaring will be performed using Gates Glidden drill #3 in a brushing motion away from dangerous zone
  Interventions: Procedure: coronal flaring
- Non coronal flaring (Active Comparator): In group B no coronal flaring will be performed following minimally invasive approach.
  Interventions: Procedure: Non coronal flaring

INTERVENTIONS:
Procedure: coronal flaring — early coronal flaring will be performed using Gates Glidden drill #3 in a brushing motion away from dangerous zone
  Arms: Early acoronal flaring
Procedure: Non coronal flaring — No coronal flaring will be performed
  Arms: Non coronal flaring

SUMMARY:
The aim of this clinical study is to evaluate the influence of early coronal flaring upon postoperative pain following root canal treatment in a single session approach.

DETAILED DESCRIPTION:
All patients will be treated in a single session approach regardless of the group. All molars will be anesthetized either through infiltration in case of maxillary molars or inferior alveolar nerve block in case of mandibular molars using Octocaine 2% with epinephrine 1: 100,000 (Lidocaine HCl, Novocol Pharmaceutical, Ontario, Canada.). Rubber dam will be applied; and access will be opened using Endo access bur.

Canals will be scouted using manual patency file in a watch winding maneuver. In group A, ProGlider PG (size 16, .02 taper) instrument with a length of 25 mm will be used to the working length, then early coronal flaring will be performed using Gates Glidden drill #3 in a brushing motion away from dangerous zone. In group B no coronal flaring will be performed following minimally invasive approach.

Root canals will be copiously irrigated using 10 ml 2.5% sodium hypochlorite NaOCl (Clorox; Egyptian Company for household bleach, Egypt) delivered using 28 Gauge safety Steri Irrigation Tip (DiaDent Group International, Burnaby, BC, Canada) inserted 3 mm below cementoenamel junction. Working length will be determined using electronic apex locator Root ZX II (J. Morita Mfg. Corp, Kyoto, Japan) and confirmed radiographically using parallel technique with receptor holding device.

Canals will be irrigated again with 10ml 1.5% NaOCl, which will be delivered 2mm coronal to apical canal terminus. Irrigation will be hydro-dynamically agitated with EndoActivator device (Dentsply Maillefer, Baillagues, Switzerland) using yellow tips #15/02 inserted 2mm short of working length for 60 seconds. ProGlider PG (size 16, .02 taper) instrument with a length of 25 mm will be used to the working length. Root canals will be shaped using ProTaper next rotary Ni-Ti files (Dentsply Maillefer, Baillagues, Switzerland) till # X3 (Elnaghy et al. 2014). Each file will be used in one molar. Finally, Root canals will be obturated using cold lateral compaction technique. The molars will be permanently restored using composite resin restoration and will be scheduled for extra coronal restoration.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient age above 18-70 years old.

  * 2. Both males and females will be included.
  * 3. All patients are in a good health without systemic condition.
  * 4. The offending tooth is a molar.
  * 5. The offending molar is indicated for root canal treatment.
  * 6. One molar for every patient.
  * 7. All patients will sign an informed consent.

Exclusion Criteria:

* 1. Necrotic molars

  * 2. The offending tooth has previous attempt of pulp therapy or root canal treatment.
  * 3. The patient showing any clinical or radiographic evidence of periapical pathosis.
  * 4. Patients received analgesics or systemic antibiotic prior to treatment.
  * 5. Immunocompromised patients.
  * 6. Any unknown infectious disease (e.g. HBV, HCV, HIV, or T.B.)
  * 7. History of cancer with radio or chemotherapy.
  * 8. Offending molar with mobility score ≥2.
  * 9. Offending molar with pocket depth ≥6mm.
  * 10. Immature molars.
  * 11. Nonodontogenic pain.
  * 12. Patients with more than one tooth requiring endodontic intervention

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | after 4hours after treatment.
  The pain level will be measured using a validated pain scale known as the Verbal Analogue scale
postoperative pain | after 6hours after treatment.
  The pain level will be measured using a validated pain scale known as the Verbal Analogue scale
postoperative pain | after 12hours after treatment.
  The pain level will be measured using a validated pain scale known as the Verbal Analogue scale
postoperative pain | after 24hours after treatment.
  The pain level will be measured using a validated pain scale known as the Verbal Analogue scale
postoperative pain | after 48 hours after treatment.
  The pain level will be measured using a validated pain scale known as the Verbal Analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Heba A ElAsfouri, Study Director — Cairo University
Locations (1):
- Cairo University Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capar ID, Arslan H, Akcay M, Ertas H. An in vitro comparison of apically extruded debris and instrumentation times with ProTaper Universal, ProTaper Next, Twisted File Adaptive, and HyFlex instruments. J Endod. 2014 Oct;40(10):1638-41. doi: 10.1016/j.joen.2014.04.004. Epub 2014 May 27. PMID 25260737